CLINICAL TRIAL: NCT01278953
Title: TactiCath Contact Force Ablation Catheter Study for Atrial Fibrillation
Acronym: TOCCASTAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VP-002 527
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-01

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: paroxysmal atrial fibrillation; atrial fibrillation; radiofrequency ablation; pulmonary vein isolation; ablation catheter; RF; contact force sensing; contact force; contact force assisted ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TactiCath (Experimental): Catheter ablation to treat paroxysmal AF using the TactiCath catheter with contact force capability
  Interventions: Device: Catheter ablation to treat paroxysmal atrial fibrillation
- Control (Active Comparator): Catheter ablation to treat paroxysmal AF using a catheter with no contact force sensing capability
  Interventions: Device: Catheter ablation to treat paroxysmal atrial fibrillation

INTERVENTIONS:
Device: Catheter ablation to treat paroxysmal atrial fibrillation — A pulmonary vein isolation procedure will be performed using radiofrequency ablation.

SUMMARY:
The TOCCASTAR Study will assess the safety and effectiveness of a contact force sensing catheter used for ablation in patients with paroxysmal atrial fibrillation. Subjects will be randomized for treatment with either the TactiCath catheter or another ablation catheter with no contact force sensing capability. Patients will be followed for 12 months to compare the incidence of serious adverse events and freedom from recurring, symptomatic AF between the two study arms. Additional measures of treatment success including quality of life, recurrence of asymptomatic AF and procedural efficiency will also be studied.

A second phase of the study will treat up to 50 non-randomized subjects with a new version of the device under the same protocol.

DETAILED DESCRIPTION:
It has been hypothesized that the ability to create durable lesions during radiofrequency (RF) ablation is directly correlated with a reduction in the recurrence of arrhythmia in patients with paroxysmal atrial fibrillation (PAF). Lesion depth is directly correlated with the contact force measured between the the tip of the catheter and the heart tissue. In this study, patients in whom a pulmonary vein isolation procedure has been prescribed for the treatment of PAF will be randomized for treatment with either a device incorporating contact force sensing or one without.

To be included in the study, patients 18 or older must demonstrate a history of atrial fibrillation and will have failed treatment using antiarrhythmic medications. In both study arms, ablation will be performed using an accepted treatment strategy and standard procedures. Patients will receive routine follow-up for 12 months after the procedure, with the addition of ambulatory monitoring to detect the recurrence of episodes of atrial arrhythmia. The study will compare the effectiveness of the procedure in the two arms, and will characterize any differences in safety outcomes primarily related to complications arising from the use of an ablation device and the ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic PAF refractory to at least one Class I-IV antiarrhythmic drug
* minimum one documented PAF episode >30 sec duration within prior 12 months
* minimum three PAF episodes during prior 12 months
* 18 years or older

Exclusion Criteria:

* persistent or long-standing persistent AF
* four or more cardioversions in prior 12 months
* MI, CABG or PCI within preceding 3 months
* left atrial diameter > 5.0 cm
* LVEF < 35%
* NYHA class III or IV
* previous left atrial ablation procedure
* previous tricuspid or mitral valve repair surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Reddy VY, Dukkipati SR, Neuzil P, Natale A, Albenque JP, Kautzner J, Shah D, Michaud G, Wharton M, Harari D, Mahapatra S, Lambert H, Mansour M. Randomized, Controlled Trial of the Safety and Effectiveness of a Contact Force-Sensing Irrigated Catheter for Ablation of Paroxysmal Atrial Fibrillation: Results of the TactiCath Contact Force Ablation Catheter Study for Atrial Fibrillation (TOCCASTAR) Study. Circulation. 2015 Sep 8;132(10):907-15. doi: 10.1161/CIRCULATIONAHA.114.014092. Epub 2015 Aug 10. PMID 26260733

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 300 subjects consented and were randomized, 5 subjects did not have the study device introduced. Thus 295 subjects contributed to study endpoints.
Groups:
- TactiCath: Ablation performed using the TactiCath contact force sensing catheter
  Catheter ablation for the treatment of paroxysmal atrial fibrillation: A pulmonary vein isolation procedure will be performed using radiofrequency ablation.
- Control: Ablation performed using a catheter with no contact force sensing capability
  Catheter ablation for the treatment of paroxysmal atrial fibrillation: A pulmonary vein isolation procedure will be performed using radiofrequency ablation.
Period: Overall Study
Arm/Group | TactiCath | Control
Started | 155 | 145
Completed | 146 | 134
Not Completed | 9 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TactiCath | Control | Total
Number analyzed (Participants) | 155 | 145 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (9.32) | 61 (10.84) | 60.3 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 54 | 109
  Male | 100 | 91 | 191
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 148 | 141 | 289
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 96 | 87 | 183
  Europe | 59 | 58 | 117

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Recurrence of Symptomatic Atrial Fibrillation, Atrial Tachycardia or Atrial Flutter
Description: Includes both acute success (successful electrical isolation of all pulmonary veins) and chronic success. Re-treatment for AF with ablation or the use of Class I or Class III antiarrhythmic drugs after a 3 month blanking period constitute a treatment failure.
Time Frame: 12 months
Population: Primary effectiveness was calculated using the Per Protocol (PP) population (n=280). 10 subjects who had PVI attempted were excluded from the PP population.due to insufficient data. A medical panel (DSMB) blinded to treatment, adjudicated the exclusion of subjects from the analysis (n=3 from TactiCath; n=7 from Control)
Measure: Number; unit: participants
Arm/Group | TactiCath | Control
Number analyzed (Participants) | 146 | 134
participants | 99 | 93

2. Primary Outcome: Incidence of Device-related Early-onset Primary Serious Adverse Events
Description: Includes serious adverse events occurring within 7 days of the index procedure or hospital discharge, whichever is later, and diagnosed at any time during the follow-up period.
Time Frame: 12 months
Population: The Safety analysis population excludes 5 subjects who signed consent and were randomized but were not exposed to the study procedure or the study device resulting in n=295 subjects. (n=3 excluded from TactiCath; n=2 excluded from the Control group)
Measure: Number; unit: participants
Arm/Group | TactiCath | Control
Number analyzed (Participants) | 152 | 143
participants | 3 | 2

ADVERSE EVENTS:
Time Frame: 12 months
Description: The Safety analysis population excludes 5 subjects who signed consent and were randomized but were not exposed to the study procedure or the study device resulting in n=295 subjects.
  3 subjects were excluded from the TactiCath group resulting in n=152 subjects 2 subjects excluded from the Control group resulting in n=143 subjects
Arm/Group | TactiCath | Control
Serious Adverse Events (participants affected / at risk) | 10/152 | 11/143
Other Adverse Events (participants affected / at risk) | 70/152 | 56/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TactiCath (N=152) | Control (N=143)
Cardiac perforation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Perforation (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Vascular Access Complication (Vascular disorders) | 3 (3) | 3 (3)
Hospitalization (General disorders) | 4 (4) | 5 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TactiCath (N=152) | Control (N=143)
Cardiac disorders (Cardiac disorders) | 38 (75) | 36 (59)
Vascular disorders (Vascular disorders) | 17 (20) | 9 (9)
Repiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 3 (3)
General disorders (General disorders) | 6 (6) | 7 (8)
Investigations (Investigations) | 6 (6) | 6 (8)
Nervous systems disorders (Nervous system disorders) | 7 (7) | 2 (4)
Gastrointestinal disorders (Gastrointestinal disorders) | 4 (4) | 4 (5)
Renal and urinary disorders (Renal and urinary disorders) | 4 (4) | 4 (4)
Infection and infestations (Infections and infestations) | 4 (4) | 2 (2)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Muskuloskeletal and connective disorders (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Eye disorders (Eye disorders) | 0 (0) | 2 (4)
Immune system disorders (Immune system disorders) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Endocrine disorders (Endocrine disorders) | 0 (0) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 0 (0) | 1 (1)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less